CLINICAL TRIAL: NCT07050147
Title: Sonographic Evaluation of Diaphragmatic Function Under Nasal High-flow (NHF) and Non-invasive Ventilation (NIV) in Respiratory Insufficiency
Acronym: SENNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Emden (Other)
Collaborators: University of Leipzig (Other)
Responsible Party: Principal Investigator, Jens Bräunlich, Clinical director, Head of department, Klinikum Emden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167/19-ek
Record Dates: First submitted 2025-01-03; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Insufficiency
Keywords: nasal high flow; NIV; diaphragm; sonography
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: This study is a randomised comparison of two investigational medical devices in a prospective, monocentric, randomised, physiological, open-label, cross-over study. Patients are randomised into two groups (study arms) with a randomisation ratio of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal high flow (Active Comparator)
  Interventions: Device: Nasal high flow
- NIV (Active Comparator)
  Interventions: Device: NIV

INTERVENTIONS:
Device: Nasal high flow — 3 sonographic measurements after use of 30 minutes
  Arms: Nasal high flow
Device: NIV — 3 sonographic measurements after 30 minutes use
  Arms: NIV

SUMMARY:
The aim of the study is to investigate the influence of respiratory support on diaphragmatic function (O2, NHF, NIV). The effects on the diaphragm, the respiratory values (FEV1, respiratory rate) and the subjective well-being of the patients during the therapy phases will be measured.

The primary objective of the clinical study is to investigate the differences in respiratory support with regard to the change in diaphragmatic kinetics and morphology (Tdi; TEx; Tdi, ee, Tdi, pi, ΔTdi, TFdi) as a function of respiratory rate.

For both ventilation modes, the influence on the respiratory situation, the respiratory muscle pump and adverse events will also be analysed. This is done using defined variables (FEV1, FEV1%VC, respiratory rate, frequency and type of adverse events (AEs), subjective satisfaction with the test product (Borg scale)).

ELIGIBILITY:
Inclusion Criteria:

* acute or chronic respiratory insufficiency with and/or hypercapnia,
* age > 18 years.
* tolerate respiratory support devices
* to sign a written declaration of consent

Exclusion Criteria:

* Presence of respiratory insufficiency requiring intubation,
* clinical instability,
* metabolic acidosis or alkalosis,
* Contraindication for NIV according to the S3 guideline,
* serious concomitant illnesses,
* unwillingness to co-operate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Sonographic measurements of diaphragm thickness | after 30 minutes use
  Tdi ee in mm = Diaphragm thickness is determined by measuring the distance between the diaphragmatic pleura and the diaphragm/peritoneum border at maximum expiration

SECONDARY OUTCOMES:
DEx | 30 minutes
  Diaphragm excursion during rest
FEV1 | 30 min
  Forced vital capacity in 1 second as % predicted
Tiffeneau - index | 30 min
  FEV1%FVC in % = definition of obstruction of the airways
Respiratory rate | 30 min
  counts the respiratory cycles in 1 minute
Tdi pi | 30 minutes
  Diaphragm thickness is determined by measuring the distance between the diaphragmatic pleura and the diaphragm/peritoneum border at maximum inspiration (Tdi, pi) in mm
TF di | 30 min
  Thickening Fraction (calculated): TFdi Diaphragm thickening fraction (change in diaphragm thickness during inspiration as a percentage [calculation from the quotient of ΔTdi and Tdi,ee])

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Yes
All data upon request
Supporting Information: Study Protocol